CLINICAL TRIAL: NCT07402902
Title: Effects of Different Caffeine Ingestion Forms on Fat Oxidation During Cycle Ergometer Exercise
Brief Title: Caffeine Strategies and Fat Oxidation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Daniel Trujillo-Colmena, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: URJC-CAF-FOX-2026
Record Dates: First submitted 2026-01-13; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fat Metabolism; Caffeine; Cycling; Exercise; Ergogenics
MeSH Terms: conditions — Motor Activity | interventions — Caffeine; Cellulose

STUDY DESIGN:
Intervention Model Description: Participants will undergo all experimental conditions (caffeine via capsule, coffee, chewing gum, and mouth rinse, and their corresponding placebos) in a randomized, double-blind, counterbalanced crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Caffeine capsule (Experimental): Participants will ingest 3 mg/kg of anhydrous caffeine powder in an opaque capsule 60 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Drug: Caffeine (Guinama Anhydrous Powder)
- Placebo capsule (Placebo Comparator): Participants will ingest an opaque capsule filled with cellulose (placebo) 60 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Other: Placebo (Cellulose Capsule)
- Caffeine coffee (Experimental): Participants will consume 3 mg/kg of caffeine via soluble coffee (Nescafé Classic) in 250 mL of hot water 60 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Dietary Supplement: Caffeine (Nescafé Classic Coffee)
- Placebo coffee (Placebo Comparator): Participants will consume decaffeinated soluble coffee (Nescafé Descafeinado) in 250 mL of hot water 60 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Other: Placebo (Decaffeinated Coffee)
- Caffeine chewing gum (Experimental): Participants will chew caffeinated gum (Kafewake) containing 3 mg/kg of caffeine for 10 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Dietary Supplement: Caffeine (Kafewake Gum)
- Placebo chewing gum (Placebo Comparator): Participants will chew non-caffeinated gum (Kafewake) with identical flavor and texture for 10 minutes before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Other: Placebo (Non-caffeine Gum)
- Caffeine mouth rinse (Experimental): Participants will perform a 20-second mouth rinse with 25 mL of water containing 3 mg/kg of caffeine from soluble coffee (Nescafé Classic) before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Other: Caffeine Mouth Rinse Solution
- Placebo mouth rinse (Placebo Comparator): Participants will perform a 20-second mouth rinse with 25 mL of water containing decaffeinated soluble coffee (Nescafé descafeinado) before performing 60 minutes of cycling on a cycle ergometer at Fatmax intensity.
  Interventions: Other: Placebo Mouth Rinse Solution

INTERVENTIONS:
Drug: Caffeine (Guinama Anhydrous Powder) — 3 mg/kg of anhydrous caffeine powder (Guinama, Spain) administered in an opaque capsule 60 min before exercise.
  Arms: Caffeine capsule
Dietary Supplement: Caffeine (Nescafé Classic Coffee) — 3 mg/kg of caffeine via Nescafé Classic (Nestlé, Switzerland) dissolved in 250 mL of water 60 min before exercise.
  Arms: Caffeine coffee
Dietary Supplement: Caffeine (Kafewake Gum) — 3 mg/kg of caffeine via Kafewake gum (Arafarma group, Spain), chewed for 10 min before exercise.
  Arms: Caffeine chewing gum
Other: Caffeine Mouth Rinse Solution — 3 mg/kg of caffeine (Nescafé Classic) dissolved in 25 mL of water for a 20-second rinse before exercise.
  Arms: Caffeine mouth rinse
Other: Placebo (Cellulose Capsule) — Opaque capsule containing cellulose powder, matching caffeine capsules, taken 60 min before exercise.
  Arms: Placebo capsule
Other: Placebo (Decaffeinated Coffee) — Decaffeinated Nescafé (Nestlé, Switzerland) in 250 mL of water, matching caffeinated coffee, taken 60 min before.
  Arms: Placebo coffee
Other: Placebo (Non-caffeine Gum) — Kafewake Non-caffeinated gum (Arafarma group, Spain) with identical taste and texture, chewed for 10 min before.
  Arms: Placebo chewing gum
Other: Placebo Mouth Rinse Solution — Decaffeinated Nescafé in 25 mL of water for a 20-second rinse immediately before exercise.
  Arms: Placebo mouth rinse

SUMMARY:
The goal of this clinical trial is to learn if different forms of caffeine ingestion can influence fat oxidation during submaximal cycling exercise. The study will recruit healthy adults, both men and women, aged 18 to 50, who regularly perform aerobic exercise. The main questions it aims to answer are:

* Does caffeine increase fat oxidation during one hour of cycling at the Fatmax intensity?
* Do different forms of caffeine ingestion (capsule, coffee, chewing gum, or mouth rinse) differ in their effect on fat oxidation?
* Do these caffeine forms alter total energy expenditure, cardiorespiratory response, or perceived exertion during exercise?
* Are there differences in the occurrence or severity of side effects between caffeine administration methods?

Researchers will compare each caffeine form to its corresponding placebo to determine their effects on fat oxidation and other physiological outcomes.

Participants will:

* Attend a pre-experimental session to determine their Fatmax intensity and VO₂max using an incremental cycling test
* Perform eight experimental sessions, each consisting of one hour of cycling at Fatmax intensity
* Receive caffeine or placebo via capsules, coffee, chewing gum, or mouth rinse according to a randomized, double-blind, crossover design
* Be monitored for fat and carbohydrate oxidation, total energy expenditure, heart rate, and perceived exertion during exercise
* Report any side effects immediately after the session and 24 hours later using a structured questionnaire

All sessions will be conducted under controlled laboratory conditions with standardized protocols to ensure safety and reliable measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-50 years
* Regular aerobic exercise at least 1 hour per day, 2 days per week
* Provide written informed consent

Exclusion Criteria:

* Smoking
* Use of medication or ergogenic supplements during the study period
* Caffeine intolerance or allergy
* Cardiopulmonary or musculoskeletal disorders
* Use of oral contraceptives in female participants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Rate of fat oxidation during submaximal cycling exercise at Fatmax intensity | 1 hour per experimental session
  Continuous measurement of fat oxidation using indirect calorimetry during 1-hour cycling at Fatmax intensity. Calculated from respiratory gas exchange (VO₂ and VCO₂) using Frayn's equations. Unit of Measure: grams per minute (g/min).

SECONDARY OUTCOMES:
Rate of carbohydrate oxidation during submaximal cycling exercise at Fatmax intensity | 1 hour per experimental session
  Continuous measurement of carbohydrate oxidation using indirect calorimetry during 1-hour cycling at Fatmax intensity. Calculated from respiratory gas exchange (VO₂ and VCO₂) using Frayn's equations. Unit of Measure: grams per minute (g/min).
Total energy expenditure during exercise | 1 hour per experimental session
  Estimated from indirect calorimetry data using Brouwer's equation, recorded continuously during 1-hour cycling at Fatmax intensity. Unit of Measure: kilocalories per minute (kcal/min).
Mean Exercise Heart Rate | 1 hour per experimental session
  Heart rate monitored continuously via a chest strap (Polar H9, Polar Electro, Findland) during the exercise test. Unit of Measure: beats per minute (bpm).
Oxygen consumption | 1 hour per experimental session
  Volume of oxygen consumed during the exercise session measured breath-by-breath via indirect calorimetry using the Ergostik gas analyzer (Geratherm Respiratory GmbH, Germany). Unit of Measure: Liters per minute (L/min).
Carbon Dioxide Production | 1 hour per experimental session
  Volume of carbon dioxide produced during the exercise session measured breath-by-breath via indirect calorimetry using the Ergostik gas analyzer (Geratherm Respiratory GmbH, Germany). Unit of Measure: Liters per minute (L/min).
Blood lactate concentration | Every 20 minutes during each 1-hour session
  Measured from capillary blood samples taken from the fingertip during exercise to assess metabolic response to different caffeine interventions. Unit of measure: Millimoles per liter (mmol/L).
Rating of Perceived Exertion (RPE) during exercise | Every 10 minutes during each 1-hour session
  Assessed using Borg's 6-20 scale; participants report perceived exertion at regular intervals. Unit of Measure: Units on a scale (from 6 to 20).
Occurrence of caffeine-related side effects | Immediately after each session and 24 hours post-exercise
  Structured questionnaire assessing symptoms commonly associated with caffeine intake, such as nervousness, tremors, insomnia, gastrointestinal discomfort, and increased heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Del Coso, PhD, Principal Investigator — Universidad Rey Juan Carlos; Arturo Casado, PhD, Principal Investigator — Universidad Rey Juan Carlos

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications may be made available upon reasonable request. These data may include anonymized metabolic, ventilatory, cardiovascular and perceptual variables collected during the study (e.g., fat oxidation rate, energy expenditure, VO₂, VCO₂, heart rate, capillary blood lactate concentration, and ratings of perceived exertion). Any data sharing will be subject to ethical approval, compliance with applicable data protection regulations, and approval by the study investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data may be shared after the publication of the main study findings and will remain available for up to three years following publication.
Access Criteria: Access to any de-identified individual participant data will be considered on a case-by-case basis. Requests will require a scientifically sound proposal and may be subject to additional ethical review and data use agreements, in accordance with institutional and legal requirements. The study investigators reserve the right to decline requests.
URL: https://www.urjc.es/contacto

REFERENCES:
- [Result] Guest NS, VanDusseldorp TA, Nelson MT, Grgic J, Schoenfeld BJ, Jenkins NDM, Arent SM, Antonio J, Stout JR, Trexler ET, Smith-Ryan AE, Goldstein ER, Kalman DS, Campbell BI. International society of sports nutrition position stand: caffeine and exercise performance. J Int Soc Sports Nutr. 2021 Jan 2;18(1):1. doi: 10.1186/s12970-020-00383-4. PMID 33388079
- [Result] Ruiz-Moreno C, Gutierrez-Hellin J, Amaro-Gahete FJ, Gonzalez-Garcia J, Giraldez-Costas V, Perez-Garcia V, Del Coso J. Caffeine increases whole-body fat oxidation during 1 h of cycling at Fatmax. Eur J Nutr. 2021 Jun;60(4):2077-2085. doi: 10.1007/s00394-020-02393-z. Epub 2020 Oct 6. PMID 33025051